CLINICAL TRIAL: NCT04265599
Title: Hypercalcemia After Cosmetic Paraffin Oil Injections: Unravelling Etiology, Pathogenesis and Potential Treatments
Brief Title: Exploring Pathogenesis and Treatment of Hypercalcemia Caused by Intramuscular Injection of Paraffinoil
Status: Recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Ebbe Eldrup, MD, DMSc, Principal investigator Consultant Endocrinologist MD DMSc, Herlev Hospital
Other Study IDs: VEK RegionH: H-19010297
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hypercalcemia; Renal Injury; Paraffinoma
MeSH Terms: conditions — Hypercalcemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples Muscle tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the study is to characterize paraffin oil induced granulomatous disease. We will investigate pathogenesis and natural history of paraffin disease. Subsequently, through further translational studies, we intend to identify novel treatments to be tested in future randomized clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* previous intramuscular injection of paraffin or other oil

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with concentration of ionized calcium in plasma above normal range = Hypercalcemia | at first examination or developed during observation period until 2025
  Hypercalcemia in plasma (exploratory not intervention study). yes or no and level.
Number of patients with concentration of parathyroid hormone PTH in plasma below normal range | at first examination or developed during observation period until 2025
  PTH level in plasma indicator of hypercalcemia

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No